CLINICAL TRIAL: NCT05908968
Title: A Pilot Study to Assess the Effects of Oxygen-enriched Water (ELO Water) on Wound Healing for Diabetic Foot Ulcers
Brief Title: Assessing the Effects of ELO Water on Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: ELO Water Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELO DFU
Record Dates: First submitted 2023-06-04; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Foot Ulcer, Diabetic
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Adults with type 2 diabetes and diabetic foot ulcer which has not healed with conventional therapy for at least 30 days prior to recruitment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drinking ELO water (Experimental): Drinking 1.5 litres of ELO water daily
  Interventions: Dietary Supplement: ELO water

INTERVENTIONS:
Dietary Supplement: ELO water — Drinking 1.5 litres daily of ELO water for 12 weeks

SUMMARY:
This pilot study examined the effects of ELO water, a commercially-available oxygen-enriched drinking water, on wound healing in patients with diabetic foot ulcers over 12 weeks.

DETAILED DESCRIPTION:
As hyperbaric chamber and topical oxygen therapies have demonstrated efficacy in improving DFU healing, the aim of this study was to evaluate ELO water, which has been shown to increase arterial oxygen levels, as a novel means of increasing oxygen delivery to poorly-healing DFUs as an adjunct to standard care. This proof-of-concept pilot study of drinking oxygen-enriched ELO water to treat diabetic foot ulcers (DFUs) was conducted on 16 adults with non-healing (for at least 30 days prior to the study) DFUs in Changi General Hospital in Singapore.

ELO water was delivered to participants' homes and their water consumption recorded in diaries, which was checked by the research co-ordinator at 2-weekly visits for 12 weeks. Minimum compliance was defined to be at least 85% of the water (12/14 bottles/fortnight), equivalent to 9 litres/week. No changes in diabetic therapy, diet or exercise were made during the study period.

All participants were seen by podiatrist for standard of care DFU treatment weekly. The ulcer size was captured following wound debridement each week using a standardized digital photographic protocol and the photos were encrypted and anonymized for confidentiality and data protection. All the images were assessed independently. Wound dressing was carried out twice per week in between visits at primary care clinics or at home.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes and haemoglobin A1c (HbA1c) at screening of 7.0-10.0% on oral glucose-lowering medication and/or insulin at a stable dose for the last three months

Exclusion Criteria:

* pregnant or lactating
* conditions which would independently worsen ulcer healing such as severe peripheral vascular disease or varicose veins
* immunosuppressive therapy
* comorbidities necessitating fluid restriction such as renal, liver or cardiac failure.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Reduction in wound area | 12 weeks
  Absolute and percentage reduction in wound area

SECONDARY OUTCOMES:
Complete wound closure | 12 weeks
  Percentage of wounds with complete closure

CONTACTS AND LOCATIONS:
Overall Officials: Joan Khoo, Principal Investigator — Changi General Hospital
Locations (1):
- Joan Khoo, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schreml S, Szeimies RM, Prantl L, Karrer S, Landthaler M, Babilas P. Oxygen in acute and chronic wound healing. Br J Dermatol. 2010 Aug;163(2):257-68. doi: 10.1111/j.1365-2133.2010.09804.x. Epub 2010 Apr 15. PMID 20394633
- [Result] Sun XK, Li R, Yang XL, Yuan L. Efficacy and safety of topical oxygen therapy for diabetic foot ulcers: An updated systematic review and meta-analysis. Int Wound J. 2022 Dec;19(8):2200-2209. doi: 10.1111/iwj.13830. Epub 2022 May 5. PMID 35510518
- [Result] Khoo J, Hagemeyer CE, Henstridge DC, Kumble S, Wang TY, Xu R, Gani L, King T, Soh SB, Puar T, Au V, Tan E, Tay TL, Kam C, Teo EK. Effects of water stably-enriched with oxygen as a novel method of tissue oxygenation on mitochondrial function, and as adjuvant therapy for type 2 diabetes in a randomized placebo-controlled trial. PLoS One. 2021 Jul 14;16(7):e0254619. doi: 10.1371/journal.pone.0254619. eCollection 2021. PMID 34260650